CLINICAL TRIAL: NCT01257243
Title: Multicentric, Randomized, Open-label Trial to Evaluate the Superiority of Fixed Dose Combination of Oxomemazine, Guaifenesin and Potassium Iodate to Guaifenesin Monotherapy in Acute Cough Treatment
Brief Title: Comparison Between Oxomemazine, Guaifenesin and Potassium Iodate Versus Guaifenesin Monotherapy in Acute Cough Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGPGEMS0110
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cough
Keywords: cough; symptoms; cold; flu
MeSH Terms: conditions — Cough; Common Cold; Influenza, Human | interventions — Guaifenesin; potassium iodate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRUG 1 (Experimental): Syrup of oxomemazine, guaifenesin and potassium iodate
  Interventions: Drug: Syrup of oxomemazine, guaifenesin and potassium iodate
- DRUG 2 (Active Comparator): Syrup of guaifenesin
  Interventions: Drug: Syrup of guaifenesin

INTERVENTIONS:
Drug: Syrup of oxomemazine, guaifenesin and potassium iodate — 5ml each 4 hours
  Arms: DRUG 1
Drug: Syrup of guaifenesin — 5ml each 4 hours
  Arms: DRUG 2

SUMMARY:
The purpose of this study is evaluate if efficacy of a combination dose of oxomemazine, guaifenesin and potassium iodate is superior than guaifenesin monotherapy in acute cough treatment.

DETAILED DESCRIPTION:
STUDY DESIGN

* Open-label, superiority, prospective, parallel group, intent to treat trial
* Experiment duration: 7 days
* 3 visits (days 1, 2 and 7)
* Reduction cough symptoms
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Patients with productive cough as result an acute URTI (i.e., cold or flu) or allergic cough in the last 10 day.
3. Cough score superior to 3.

Exclusion Criteria:

1. Pregnancy or risk of pregnancy.
2. Lactation.
3. Fever above 38º C.
4. Patients with bacterial infections of the upper respiratory tract.
5. Any pathology or past medical condition that can interfere with this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-10-25 (Actual)

PRIMARY OUTCOMES:
Reduction/improvement of cough symptoms | DAY 7
  The reduction of cough symptoms will be evaluated by comparative score index basal and final score

SECONDARY OUTCOMES:
Tolerance | DAY 7
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Pinho, MD, Study Director — EMS
Locations (1):
- Beneficência Nipo Brasileira de São Paulo - Hospital Nipo Brasileiro, São Paulo, Brazil